CLINICAL TRIAL: NCT06979167
Title: Study on Complications After Midline Catheter Placement and the Risk Factors in Children
Brief Title: Complications of Midline Catheter in Surgical Children
Acronym: MIDline
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Other Study IDs: 2503-174-1626
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Midline Catheter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- midline catheter inserted group
  Interventions: Device: midline catheter insertion during general anesthesia

INTERVENTIONS:
Device: midline catheter insertion during general anesthesia — This intervention involves the ultrasound-guided insertion of a midline catheter into a peripheral vein (basilic, cephalic, or brachial vein) during general anesthesia in pediatric patients.

SUMMARY:
The goal of this observational study is to understand the incidence and risk factors of complications associated with midline catheter placement in pediatric patients (under 18 years old) undergoing general anesthesia. The main questions it aims to answer are:

What is the overall complication rate (including malfunction, bleeding, thrombosis, inflammation, and infection) after midline catheter placement in children?

What factors (e.g., age, weight, vein diameter, insertion site, catheter maintenance duration) are associated with a higher risk of complications?

Participants will:

Receive a midline catheter during surgery under general anesthesia.

Undergo ultrasound-guided assessment of the catheter site immediately after placement, 24 hours later, and before the catheter is removed.

Be monitored for any complications related to the catheter, including infection, blood clots, or blockage.

This study will help identify which factors increase the risk of complications, improving the safe use of midline catheters in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients under 18 years of age
* Scheduled to undergo general anesthesia for surgery at Seoul National University Children's Hospital.
* Clinically indicated for midline catheter insertion as determined by the attending anesthesiologist.

Exclusion Criteria:

* Patients requiring central venous catheter (CVC) insertion instead of a midline catheter.
* Known coagulation disorders.
* History of severe thrombosis.
* Any other conditions that, in the investigator's judgment, make the patient unsuitable for the study.

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study will include pediatric patients under 18 years of age who are undergoing general anesthesia for surgery at Seoul National University Hospital and require midline catheter placement. This population is selected to investigate the incidence and risk factors for complications associated with midline catheter insertion in pediatric patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2028-02-25 (Estimated); Study Completion 2028-03-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Complications Related to Midline Catheter | From midline catheter insertion to catheter removal (up to 7 days).
  The overall complication rate is defined as the proportion of patients experiencing any catheter-related complications, including catheter malfunction, infection (clinical signs or positive culture), bleeding at the insertion site, thrombosis (confirmed by ultrasound), and catheter dislodgement.

SECONDARY OUTCOMES:
Number of Participants with Each Type of Complication | From midline catheter insertion to catheter removal (up to 7 days).
  The incidence of each specific complication type will be recorded, including:
  Catheter malfunction (clinical assessment), Infection (clinical signs or positive culture), Bleeding at the insertion site (visual inspection), Thrombosis (confirmed by ultrasound), Catheter dislodgement (clinical assessment)
Midline Catheter Maintenance Duration | From midline catheter insertion to catheter removal (up to 7 days).
  The total duration (in days) that each patient maintains a functional midline catheter without premature removal.
Number of Participants with Premature Catheter Removal and Reasons | From midline catheter insertion to catheter removal (up to 7 days).
  The primary reason for catheter removal will be documented, including: Planned removal (completion of clinical need), Premature removal due to complications (infection, malfunction, thrombosis, or patient discomfort)
Number of Participants with Thrombosis Confirmed by Ultrasound | From midline catheter insertion to catheter removal (up to 7 days)
  The presence of thrombosis at the catheter site will be assessed using ultrasound. Ultrasound will be performed immediately after insertion, 24 hours later, and at the time of catheter removal. Thrombosis will be defined as the presence of an intraluminal thrombus or significant vein narrowing.
Number of participants receiving treatment for Complications | From midline catheter insertion to catheter removal (up to 7 days)
  This outcome measures the frequency and types of treatments administered for complications associated with the midline catheter, including:
  * Antibiotics for infection (based on clinical signs or positive culture).
  * Anticoagulants for thrombosis (confirmed by ultrasound).
  * Additional catheter procedures (replacement, adjustment, or removal).
  * Analgesics or anti-inflammatory medications for local inflammation or pain. Each treatment will be documented, including the type, dose, route, and reason for administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Children's Hospital, Seoul, Seoul, South Korea